CLINICAL TRIAL: NCT06587243
Title: "Facts Tell… and With Stories Sell?" Combining Viewer-tailored Personal HPV Narrative Video With HPV Vaccine Information Video to Improve HPV Vaccine Uptake
Brief Title: "Facts Tell… and With Stories Sell?" Combining Viewer-tailored Personal Human Papillomavirus (HPV) Narrative Video With HPV Vaccine Information Video to Improve HPV Vaccine Uptake
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00030227
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Vaccination
Keywords: HPV; Vaccine; Narrative; Communication; Videos
MeSH Terms: conditions — Narration; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control (No Intervention): No videos
- Animation Only (Experimental): informational animation video only
  Interventions: Behavioral: Informational Animation Video
- Narrative Only (Experimental): personal narrative video only
  Interventions: Behavioral: Personal Narrative Video
- Narrative Then Animation (Experimental): personal narrative video followed immediately by the informational animation video
  Interventions: Behavioral: Informational Animation Video; Behavioral: Personal Narrative Video
- Animation Then Narrative (Experimental): informational animation video followed immediately by the personal narrative video
  Interventions: Behavioral: Informational Animation Video; Behavioral: Personal Narrative Video

INTERVENTIONS:
Behavioral: Informational Animation Video — The informational animation video will also take several minutes and will cover HPV disease, address specific concerns when identified, and the importance and safety of HPV vaccines.
  Arms: Animation Only; Animation Then Narrative; Narrative Then Animation
Behavioral: Personal Narrative Video — Personal narrative videos will consist of someone describing the person's own personal experience with HPV. The investigators have a collection of videos of personal narratives from different people that the investigators have cut to approximate several minutes in length so the investigators can tailor the personal narratives to match each study participant's race/ethnicity and gender as closely as possible.
  Arms: Animation Then Narrative; Narrative Only; Narrative Then Animation

SUMMARY:
This study will compare the use of informational videos only, personal story videos only, and the combination of both, to see which is most effective in increasing HPV vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Parents of 11-17 year olds not yet vaccinated against HPV

Exclusion Criteria:

* Parents whose adolescent children are already vaccinated against HPV
* Participants who do not complete the survey
* Participants who are unable or refuse to view and listen to videos on the participant's device

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who receive HPV vaccination | 9-month follow-up
  HPV vaccination will be a binary variable (received vs not received)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Salmon, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Ipsos, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No